CLINICAL TRIAL: NCT00736710
Title: Effects of rTMS on Smoking Cessation and Cognitive Outcomes in Outpatients With Schizophrenia Treated With Transdermal Nicotine Patch
Brief Title: rTMS Effects on Smoking Cessation and Cognition in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Tony George, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 121/2007
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Cigarette Smoking; Schizophrenia
Keywords: Repetitive Transcranial Magnetic Stimulation; Cigarette smoking; Schizophrenia; Randomized; Double-blind; Placebo-controlled; longitudinal; nicotine patch
MeSH Terms: conditions — Cigarette Smoking; Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)
- 2 (Sham Comparator)
  Interventions: Procedure: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS) — The rTMS procedures will be delivered in a single-blind fashion by the rTMS technician at the CAMH rTMS Laboratory. All subjects would be enrolled in a 10-week smoking cessation program using weekly group behavioral therapy which will emphasize psychoeducation about the effects of smoking on psychiatric and medical aspects of schizophrenia, social skills training, relapse-prevention skills training and benefits of quitting smoking. All subjects would start group therapy interventions in Week 1 of the trial, and begin rTMS procedures in a separate session on Week 2. The transdermal nicotine patch (TNP; 21 mg/24h) would be applied during the quit date at Week 3 (Day 15). At the end of the 10-week trial, TNP and group therapy would be discontinued.
  Arms: 1
Procedure: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — The rTMS procedures will be delivered in a single-blind fashion by the rTMS technician at the CAMH rTMS Laboratory. All subjects would be enrolled in a 10-week smoking cessation program using weekly group behavioral therapy which will emphasize psychoeducation about the effects of smoking on psychiatric and medical aspects of schizophrenia, social skills training, relapse-prevention skills training and benefits of quitting smoking. All subjects would start group therapy interventions in Week 1 of the trial, and begin rTMS procedures in a separate session on Week 2. The transdermal nicotine patch (TNP; 21 mg/24h) would be applied during the quit date at Week 3 (Day 15). At the end of the 10-week trial, TNP and group therapy would be discontinued.
  Arms: 2

SUMMARY:
Patients with schizophrenia have high rates of cigarette smoking and tobacco dependence, and great difficulties in quitting smoking. The development of novel and more effective treatments for tobacco dependence in this population is thus needed. This study will test the hypothesis that repetitive transcranial magnetic stimulation (rTMS) may facilitate smoking cessation with the transdermal nicotine patch (TNP) in patients with schizophrenia motivated to quit smoking. A total of N=40 smokers with schizophrenia would be assigned to either active rTMS (N=20) or sham rTMS (N=20) as a treatment regimen of 5X/week treatments for four weeks. All subjects would receive TNP (21 mg/24h) and weekly group behavioral therapy for smoking cessation for a total of 10 weeks. The investigators predict that active rTMS will be well-tolerated and superior to sham rTMS for enhancing smoking cessation rates in smokers with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Smoking at least 10 cigarettes per day and a Fagerstrom score of at least 4.
* Willing to quit smoking in the next 30 days.

Exclusion Criteria:

* Active alcohol or illicit drug abuse or dependence in the past 3 months
* A history of seizures, head trauma or space occupying lesions.
* A history of alcohol or illicit drug abuse in the past 6 months.
* Intolerance of the nicotine patch or its excipients
* Evidence for psychiatric instability as judged by acute psychotic exacerbations, suicidal or homicidal ideation.
* Females who are pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence (7-day point prevalence) at trial endpoint (Days 63-70) as assessed by self-reported smoking abstinence plus Expired Breath Carbon Monoxide Level <10ppm. | trial endpoint

SECONDARY OUTCOMES:
P50/NI, N-Back and VSWM Working Memory Performance | intermittent
Expired Breath Carbon Monoxide Levels | intermittent
Tobacco Craving (Tiffany QSU) and Withdrawal (Minnesota NMS) | intemittent

CONTACTS AND LOCATIONS:
Overall Officials: Tony George, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kozak K, Sharif-Razi M, Morozova M, Gaudette EV, Barr MS, Daskalakis ZJ, Blumberger DM, George TP. Effects of short-term, high-frequency repetitive transcranial magnetic stimulation to bilateral dorsolateral prefrontal cortex on smoking behavior and cognition in patients with schizophrenia and non-psychiatric controls. Schizophr Res. 2018 Jul;197:441-443. doi: 10.1016/j.schres.2018.02.015. Epub 2018 Feb 24. PMID 29486960
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research